CLINICAL TRIAL: NCT02936466
Title: Evaluation of a Serious Game for Patients With Bipolar Disorder Involved in a Psychoeducation Group
Acronym: Bipolife
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties encountered in recruiting and stop of funding
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF 9238; 2013-A01481-44 (Other: Agence Nationale de Sécurité des Médicaments)
Record Dates: First submitted 2016-07-15; First posted 2016-10-18 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Bipolar Disorders; Euthymic Status
Keywords: Psychiatry; Randomized controlled trial; Bipolar disorder; Serious game; Compliance; Psychoeducation
MeSH Terms: conditions — Bipolar Disorder; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional group (Experimental): Bipolife group
  Interventions: Behavioral: Bipolife® group
- Control group (No Intervention): No specific intervention, treatment as usual

INTERVENTIONS:
Behavioral: Bipolife® group — The participant is proposed to play to the serious game Bipolife® with following instructions :
  * At least one connection per week during 4 weeks
  * Connection time is free On add on of usual treatment After the 4 weeks and the first visit (V1), the participant can continue to participate to the serious game as much as he wishes, without any specific instructions.
  After connecting to the site www.bipolar.ubi.com, the participant is proposed to create his avatar and conduct him on his house. He realizes different kind of daily actions (like sleeping, sport activity, cooking) ; every action lead to win or to loose "energy" and "mood" points. The final aim is to stabilize the avatar's mood. Thanks to this experience, the participant can learn to distinguish positive and negative actions impacting on his condition.
  Arms: Interventional group

SUMMARY:
Bipolar disorder is a condition characterized by succession of episodes- manic, hypomanic, and depressive episodes. Major risks factors of relapses are poor compliance, sleep disorder, and toxics consumption. The aims of psychoeducation programs are to increase compliance and knowledge about bipolar disorder. Serious game are supposed, in bipolar disorder, to strengthen the efficacy of psychoeducation programs. Bipolife® is a serious game which purpose is to help bipolar patients to deal with their conditions, through 3 mains messages : to pursue the treatment, to have daily routine and to request the psychiatrist in case of relapse.

This is a multicentric randomized controlled study with two harms parallels. After a classic psychoeducation group program, patients are randomized in two groups : interventional group and control group with treatment as usual.

The main objective is to evaluate the observance in the two groups. The other objectives are to evaluate daily routine, global functioning, and access to health care. Evaluations are realized at one and four months after inclusion visit. Acceptability and satisfaction about the serious game Bipolife® will be assessed in the interventional group.

DETAILED DESCRIPTION:
Bipolife® is a serious game for bipolar patients, developed by Astra Zeneca laboratory in collaboration with a french company named Ubisoft. The aim of this interactive tool is to help patient to have a better understanding of their condition and to identify their daily routine which can impact on it.

Three visits :

At the inclusion visit (V0), on the 15days following the end of the psychoeducation group, the investigator evaluate mood, habits, daily routine, and verify inclusion criteria of the participants, in particular euthymic status. The participants are randomized by bloc in each center, in two groups : interventional group (Bipolife®) and control group.

Instructions on interventional group are to periodically connect to BIPOLIFE until next visit.

On the first visit, one month later (V1) and on the second visit, four months later (V2), the investigator evaluate compliance, routine habits and mood.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of bipolar disorder according to the Diagnostic and Statistical Manual (DSM) IV
* euthymic status at least since 3 months
* participation to a psychoeducation group ending on the 15 last days
* realized at less 50% of the sessions of psychoeducation group
* free access to a computer with internet connection
* signed informed consent

Exclusion criteria:

* decline of participation
* patient on protective measures (guardianship or trusteeship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
Compliance rate | At 4 months after the inclusion
  Evaluation of patient compliance by Medication Adherence Rating Scale (MARS) score.

SECONDARY OUTCOMES:
Evolution of toxic consumption | Between 1 and 4 months after the inclusion
  evaluation of toxic consumption : patient will be asked about his consumption, and to pass the french scale Cut-down, Annoyed, Guilty, Eye-opener (CAGE- DETA)
Evolution of sleep disturbance | Between 1 and 4 months after the inclusion
  evaluation of sleep disturbance (by Pittsburgh Sleep Quality Index PSQI)
Evolution of the alimentation | Between 1 and 4 months after the inclusion
  evaluation of alimentation (patient will be asked about his alimentation)
Global functioning | At 1 and 4 months after the inclusion
  evaluation of global functioning is realized by the Functioning Assessment Short Test (FAST) scale.
Ability to access health care in emergency description : number of emergency consultation for psychiatric reason | At 1 and 4 months after the inclusion
  evaluation of the ability to require to health care structures : Patients will be asked about their consultations and hospitalisations during the follow-up
acceptability and satisfaction | At 1 and 4 months after the inclusion
  only on the "interventional group" : evaluation of the acceptability and satisfaction by a home made acceptability scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University Montpellier Hospital, Montpellier, France